CLINICAL TRIAL: NCT03622541
Title: Using Sorafenib as a Salvage Treatment for Relapsed or Refractory Acute Myeloid Leukemia Carrying FLT3 Internal Tandem Duplication (ITD)
Brief Title: Using Sorafenib as a Salvage Treatment for Relapsed or Refractory Acute Myeloid Leukemia Carrying FLT3-ITD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Anskar Y.H. Leung, clinical professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML004
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: FLT3-ITD Mutation; AML
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sorafenib (Experimental)
  Interventions: Drug: Sorafenib 200mg

INTERVENTIONS:
Drug: Sorafenib 200mg — Sorafenib is a multi-kinase inhibitor which is FDA approved for the treatment of metastatic hepatocellular and renal cell carcinomas.
  Other Names: Sorafenib

SUMMARY:
Patients with refractory or relapsed acute myeloid leukemia (AML) after two courses of standard chemotherapy regimens have very limited options. Further chemotherapy is associated with significant toxicity and is generally ineffective. About 10-30% patients with AML carry a gain-of-function mutation of a gene known as Flt3 in the leukemic cells, conferring them with abnormal cellular proliferation. Sorafenib is a multi-kinase inhibitor which was licensed in Hong Kong for the treatment of advanced hepatocellular and renal cell carcinoma. The drug has also been shown to be effective against Flt3 and AML but it has not been licensed for use in this condition.

DETAILED DESCRIPTION:
AML is one of the most lethal cancers among young people in Hong Kong. Induction chemotherapy is the mainstay of treatment, resulting in remission (i.e. clearance of leukemic cells) in 70% cases. Patients who fail induction chemotherapy or who relapse after initial remission would need to receive further chemotherapy with a view to achieve a second remission. Those who do so can be potentially cured by bone marrow transplantation (BMT). Those who fail are left with very little options. As a result, only 30% patients can survive long-term.

AML is heterogeneous and 10-30% patients carry a gain-of-function mutation of a gene known as fms-related tyrosine kinase-3 (Flt3) in the leukemic cells, which confers them with abnormal cellular proliferation. These patients have inferior prognosis compared with those without the mutation. With conventional chemotherapy, these leukemias often fail to remit, precluding patients from receiving curative BMT. Sorafenib is a multi-kinase inhibitor which is FDA approved for the treatment of metastatic hepatocellular and renal cell carcinomas. It is also effective against Flt3 and has been shown to be very effective in inducing remission in patients with AML carrying Flt3 mutation.

This proposal aims to treat relapsed or refractory AML patients carrying Flt3 mutation in the following ways:

1. Patients who have persistent or refractory leukemia after at least two prior chemotherapy regimens will receive sorafenib to induce a remission, hence bridging them to BMT for curative treatment.
2. Patients who relapse after BMT will receive sorafenib to induce remission again in preparation for second BMT.
3. Patients who are not candidates for BMT but have persistent or refractory leukemia after at least two prior chemotherapy regimens will receive sorafenib to induce a remission, followed by chemotherapy consolidation. Sorafenib induction will have significantly less side-effects compared with induction by conventional chemotherapy.

Patients who are treated with sorafenib will be managed in the hospital and out-patient clinics in the same way as patients undergoing induction by conventional chemotherapy. They will have bone marrow examinations before and one month after receiving sorafenib treatment

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with AML carrying Flt3 mutation; AND,
* 2. Patients with persistent leukemia despite at least two prior chemotherapy regimens

Exclusion Criteria:

* Patients who are considered not fit for any form of leukemia treatment by the attending hematologists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-11-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR): | up to 16 weeks
  count ≥ 100 x109/L.

CONTACTS AND LOCATIONS:
Overall Officials: Anskar Leung, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No